CLINICAL TRIAL: NCT01904916
Title: Protocol to Obtain Tumor Biopsies From Patients With Locally Advanced (Incurable) or Metastatic Cancer to Improve Selection for Clinical Trials. (CPCT - 05 Biopsy Protocol Patient Selection)
Brief Title: CPCT-05 Biopsy Protocol Patient Selection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: P.O. Witteveen (Other)
Collaborators: The Netherlands Cancer Institute (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor-Investigator, P.O. Witteveen, Investigator, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL.45677.041.13
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Solid Tumors; Metastatic Disease
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Histological biopsy procedure (Other): This is a diagnostic multicenter study combining histological biopsy of tumor material with DNA sequencing using Ion Torrent®, Next Generation Sequencing (NGS) platform. The study aims improve stratification of cancer patients by obtaining fresh tumor biopsies for next-generation sequencing for participation in clinical trials.
  Interventions: Procedure: Histological biopsy procedure

INTERVENTIONS:
Procedure: Histological biopsy procedure

SUMMARY:
Our knowledge on the genetic mutations in cancer is rapidly expanding and we are increasingly testing drugs in mainly metastatic cancer patient populations with rare mutations. Successful examples of this new strategy are ALK inhibitors in ALK translocated NSCLC (less than 5% frequency) and EGFR inhibitors in EGFR mutant NSCLC (approximately 5% frequency). Selecting molecularly stratified patient populations for studies benefits the patient as it increases the odds of obtaining benefit from experimental treatment, especially in early clinical trials. Moreover it increases the speed and efficacy of drug development as signs of efficacy are picked up in earlier phases. Therefore, broad screening of molecular lesions in the tumors of patients that are being considered for participation in trials is crucial. This pre-selection increases our ability to perform several trials in parallel and thus include more patients in more meaningful trials. With the still dismal prognosis of patients with metastatic cancer, increasing the accrual rate to pivotal trials in selected patient populations is a key factor in improving prognosis.

The advent of Next Generation Sequencing (NGS) platforms enables us to probe a limited number of cancer related genes within 2-4 weeks. We have extensively piloted this approach and are now able to deliver clinically meaningful turn-around-times. This development enables us to use this technology to enrich clinical trials using targeted therapies for patients with specific mutations.

We will obtain tumor biopsies of a metastatic or locally advanced lesion and a peripheral blood sample from all patients included in the trial; the biopsies to obtain information on the tumor related genetic mutations (mutational profile) and the blood samples to assess each patient's germline DNA background variation. As patients will be asked to undergo an invasive procedure it is important to address the potential safety issues. Review of the literature and our own experience show that tumor biopsies can be performed with only minor complications and acceptable risks. We will recruit patients with metastatic or locally advanced solid tumors from patients that can potentially be included in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced (incurable) or metastatic cancer from a histological or cytological proven solid tumor
* Indication for systemic treatment with anti-cancer agents (with no treatment options with curative intent)
* Measurable locally advanced (incurable) or metastatic lesion(s), according to RECIST 1.1 criteria.
* Safe biopsy of a metastatic or locally advanced lesion possible
* No contraindications for lidocaine (or its derivatives) and/or midazolam and/or phentanyl
* Adequate organ function
* WHO performance status 0-2
* Age > 18 yr
* Expected adequacy to follow up
* Written informed consent

Exclusion Criteria:

• If one or more of the above mentioned inclusion criteria is not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Percentage of screened patients allocated to trials based upon outcome of genetic screening effort. | 1 year

SECONDARY OUTCOMES:
Number and nature of (serious) adverse events of the performed histological biopsies. | 2 days after each biopsy procedure
Number of samples stored for future related research. | 1 year
Number of samples with an adequate microRNA, (phospho)proteomic profiles and organoid cultures that allows biomarker discovery efforts. These profiles will be deposited in the CPCT database. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Langenberg, MD, PhD, Principal Investigator — UMC Utrecht; Neeltje Steeghs, MD, PhD, Principal Investigator — Antoni van Leeuwenhoek Hospital; Maja J.A. de Jonge, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (3):
- Netherlands (3):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht